CLINICAL TRIAL: NCT01718236
Title: Modern Myorelaxation Procedure and Reversal of Neuromuscular Blockade With General Anesthesia for Caesarean Section
Acronym: RocSugIO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brno University Hospital (Other)
Collaborators: St. Anne's University Hospital Brno, Czech Republic (Other); University Hospital Olomouc (Other); IGA - internal grant agency, Ministry of Health (Unknown)
Responsible Party: Principal Investigator, Petr Štourač, MD, MD, Brno University Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IGA NT 13906-4
Record Dates: First submitted 2012-10-24; First posted 2012-10-31 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Caesarean Section; Pregnancy
Keywords: caesarean section; rocuronium; sugammadex
MeSH Terms: interventions — Rocuronium; Sugammadex; Succinylcholine; Neostigmine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rocuronium + sugammadex (Experimental): Intubation after rocuronium administration and reversal of blockade after administration of sugammadex
  Interventions: Drug: Rocuronium + sugammadex
- Succinylcholine + Neostigmine (Experimental): Intubation after succinylcholine administration, neuromuscular block is than maintained by rocuronium administration and reversal of block is by neostigmine + atropine administration
  Interventions: Drug: Succinylcholine + Neostigmine

INTERVENTIONS:
Drug: Rocuronium + sugammadex — Administration of rocuronium 1 mg/kg, intubation at decrease in Single Twitch to 10% of baseline event. by the disappearance of visible spikes event. in the 60th seconds after administration of muscle relaxants. Anesthesia with sevoflurane according to the MAC, neuromuscular blockade TOF count at 1-2.At the end of operation at PTC 1-2 sugammadex 4 mg/kg, at the TOF count 1-2, sugammadex 2 mg/kg, in the case of failure to achieve these values the anesthesiologist will wait until the minimum value of PTC 1-2 will be achieved. In can not intubate can not ventilate, and the failure of the introduction of laryngeal masks sugammadex 16mg/kg, immediately following the discovery of this fact and wait for the recovery of muscle strength. Time to recovery is recorded.
  Arms: Rocuronium + sugammadex
Drug: Succinylcholine + Neostigmine — 1mg/kg succinylcholine iodide, intubation after decrease in Single Twitch to 10% of baseline event. after the disappearance of visible fasciculation event. in the 60th seconds after administration of muscle relaxants. Anesthesia with sevoflurane according to the MAC, at the moment of 20-30% of the original value of Single Twitch rocuronium 0.3 mg / kg, maintaining TOF Count at 1-2.At the end of operation at TOF Count 1-2 atropine 0.01 mg/kg and neostigmine 0.03 mg/kg. If TOF not 1-2 wait.In can not intubate can not ventilate, wait for the spontaneous recovery. Time to recovery of muscle strength is recorded.
  Arms: Succinylcholine + Neostigmine

SUMMARY:
The project aims to introduce into clinical practice for Caesarean section conducted under general anesthesia with the rapid induction myorelaxation with rocuronium and the reversal of neuromuscular blockade by using sugammadex. The aim is to demonstrate at least the same efficiency and confirm the safety of the procedure for both mother and newborn compared with older procedure.

DETAILED DESCRIPTION:
Project "Modern myorelaxation procedure and reversal of neuromuscular blockade during general anesthesia for caesarean section" aims to introduce in other indications for rapid induction of general anesthesia common and safe, alternative method of combining short-acting intravenous anesthetics propofol and fast-onset non-depolarizing muscle relaxant rocuronium into the clinical practice and demonstrate the efficacy and safety in this indication. At the same time to demonstrate the benefits of using modern reversal of neuromuscular blockade by sugammadex in termination the caesarean section under general anesthesia. Both procedures will be monitored by clinical observation, monitoring instrumentation and laboratory examination of mother and fetus (newborn) in various stages of peripartal period. The main benefit of this procedure will be in particular risk groups of mothers which are indicated by Caesarean Section while neuraxial blockade is contraindicated.

ELIGIBILITY:
Inclusion Criteria:

* caesarian section under general anesthesia in informed patient (after interview with anesthesiologist and obtain the signature for informed consent)

Exclusion Criteria:

* patient disagreement
* indicated and performed neuraxial blockade
* the anesthesiologist or obstetrician opposition to their inclusion in the study
* allergy or intolerance to one or more of study drug or known allergies or reactions to iodine

Ages: 14 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2012-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
time needed to tracheal intubation | 2 years
  Quality: Rapid induction to general anesthesia with administration propofol and rocuronium for termination the pregnancy by Caesarean section are at least as good as the combination of propofol and succinylcholine iodide.Recording and evaluated will be the time from the beginning as the first drug in the rapid induction to general anesthesia will be administered until the discovery of the first wave of etCO2 after successful intubation (seconds), evaluation of intubation conditions (resistance to laryngoscopy, position of the vocal cords, response to the intubation attempt (limbs movement or cough) scored 1-3 according to level terms, conditions, entry scores for direct visualization of the vocal cords by Cormack-Lehane (I-IV)

SECONDARY OUTCOMES:
total procedure time | 2 years
  Economics: After reversal of neuromuscular blockade using sugammadex are procedure time and turnovers shorter than the use of neostigmine in the recommended dosage for patients undergoing termination of pregnancy by Caesarean section. Recording and evaluated will be the total procedure time until the recovery from neuromuscular blockade to the level of TOF ratio of 0.9, the administration of the recovery dose will in group ROCSUG in the case for posttetanic count mode in the level of PTC1, 2 at a dose of sugammadex 4mg/kg , the TOF count 1.2 sugammadex at a dose of 2 mg / kg, in the case of failure to achieve these values the anesthesiologist wil wait with the administration of the recovery dose for their achievement. In group SUCNEO for achieving TOF count 1.2 and higher, the dose of atropine to 0.01 mg / kg and neostigmine 0.03 mg / kg will be administered.

OTHER OUTCOMES:
complications during anesthesia and during perioperation period | 2 years
  Rocuronium, sugammadex doesn´t lead to the deterioration of perinatal parameters and leads to fewer complications during anesthesia and postoperative period against a combination of succinylcholine iodide, rocuronium and neostigmine.Demographic characteristics (age,weight,BMI,gain in pregnancy,previous pregnancy, complications during pregnancy,medication during pregnancy), multiple gestation,parity,fetal position,the reason for the indication of caesarean section, the reason for general anesthesia caesarean section,week of termination of pregnancy,fetal weight,umbilical cord blood pH, pCO2,pO2,BE,Apgar,sex of the fetus,STAN or CTG assessment,the nature of amniotic fluid,time to cutting the umbilical cord will be monitored. Anesthesia complications (present or absent),the evaluation questionnaire of subjective feelings of the patient 1 day after caesarean section - sore throat,vigilance during anesthesia,myalgia,diplopia,weakness,inability to cough,shortness of breath will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, MD, Study Director — Brno Faculty hospital, department of anesthesiology and intensive care medicine
Locations (2):
- Czechia (2):
  - Faculty Hospital Olomouc, Olomouc, Olomoucký kraj
  - Faculty hospital Brno, Brno, South Moravian

REFERENCES:
- See also: Published results of the study, full text available by principal investigator Stourac Petr.MD.Ph.D Doc. — http://journals.lww.com/anesthesia-analgesia/Abstract/2016/05000/Low_Dose_or_High_Dose_Rocuronium_Reversed_with.43.aspx